CLINICAL TRIAL: NCT06837428
Title: Peer Comparison-based Risk Communication (PRICOM): A Study Protocol to Evaluate the Feasibility of Delivering a Risk Communication Intervention in the Primary Care Setting for Adults With Type 2 Diabetes Mellitus
Brief Title: Peer Comparison-based Risk Communication
Acronym: PRICOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SingHealth Polyclinics (Other)
Responsible Party: Principal Investigator, Ong Ruiheng, Principal Investigator, SingHealth Polyclinics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-2306
Record Dates: First submitted 2021-10-06; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention group will attend a risk communication session delivered by the study team and will receive a diabetes pamphlet. This estimated to take 10-15 minutes and will be back-to-back with the patient's routine clinic appointment.
  Interventions: Other: Peer comparison-based Risk Communication (PRICOM)
- Control (No Intervention): The control group will receive a diabetes pamphlet at their routine clinic appointment but will not attend a PRICOM session.

INTERVENTIONS:
Other: Peer comparison-based Risk Communication (PRICOM) — Based on the Health Belief Model, a risk communication intervention, Peer comparison-based Risk Communication (PRICOM), was developed for primary care physicians to counsel patients with T2DM on their glycaemic control and the complications that could arise, and to recommend ways to improve glycaemic control and prevent complications (or further complications). This will be supported by information from an AI (Artificial Intelligence) based diabetes tool. PRICOM aims to promote health actions in patients with T2DM by increasing their risk perceptions of diabetes complications.
  Arms: Intervention

SUMMARY:
The study objective is to evaluate the feasibility of delivering a risk communication intervention, Peer comparison-based Risk Communication (PRICOM), in the primary care setting for adults with poor T2DM control. Findings from the study will inform further revisions to PRICOM and provide an estimated effect size to estimate the required sample size for a multi-site trial.

DETAILED DESCRIPTION:
Background: Younger adults with Type 2 Diabetes Mellitus (T2DM) in Singapore tend to have poorer glycaemic control and medication adherence, factors correlating with high risk of diabetes complications. Late-stage diabetes and its complications are perceived to be slow-progressing and not immediately life-threatening. These reflect a concerning state of diabetes control and risk perception in Singapore. Using the Health Belief Model, a risk communication intervention, Peer comparison-based Risk Communication (PRICOM), was developed for physicians to counsel patients with T2DM supported by a digital tool. PRICOM aims to promote health actions by increasing their risk perceptions of diabetes complications.

Specific aims: The primary aim is to evaluate the feasibility of delivering PRICOM in the primary care setting for adults with poor T2DM control - in terms of recruitment, retention, PRICOM adherence, estimated effect size of score changes in risk perception, health actions and HbA1c change. Secondary aims are to assess validity of the risk perception scale, and to explore patients' perspectives of PRICOM.

Methodology: A multi-site randomised controlled trial will be conducted at a primary care clinic in 2 concurrent phases. In phase 1, content validation and test-retest reliability of a risk perception scale will be carried out. In phase 2, a two-arm randomised controlled trial will be conducted using mixed-methods to evaluate the feasibility of delivering PRICOM. A total 40 patient participants will be recruited by convenience sampling. Eligible patients must be age 40-79 years and have poor T2DM control with at least one HbA1c reading ≥ 8.0% within the last 6 months.

Relevance/significance of the study: Findings from the study will inform further revisions to PRICOM and provide an estimated effect size to estimate the required sample size for a multi-site trial.

ELIGIBILITY:
Eligibility criteria for patient participation:

* T2DM on follow-up at the respective study site for at least 12 months
* Age 40 to 79 years
* At least one HbA1c reading ≥ 8.0% within the last 6 months
* Able to read and speak English

Exclusion criteria for patient participation:

* Not a Singapore citizen or permanent resident
* Pregnant
* End-stage kidney disease or on renal replacement therapy
* Known terminal illness
* Visual and/or hearing impairment
* Cognitive impairment or mental illness
* Unable to provide informed consent

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Risk perception score change | 6 months
  Score change of RPS-DM (Risk Perception Scale - Diabetes Mellitus) questionnaire
Recruitment rate | 6 months
  % patients eligible to participate who were recruited
Retention rate | 6 months
  % patient participants who completed the study

SECONDARY OUTCOMES:
Self-care activity score change | 6 months
  Score change of SDSCA (Summary of Diabetes Self-Care Activities) questionnaire
Medication adherence score change | 6 months
  Score change of MARS-5 (5-item Medication Adherence Report Scale) questionnaire
HbA1c change | 6 months
  Change in HbA1c value
Perspectives of PRICOM | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ruiheng Ong, Principal Investigator — SingHealth Polyclinics
Locations (1):
- SingHealth Polyclinics - Bedok Polyclinic, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication

REFERENCES:
- [Background] Png ME, Yoong J, Phan TP, Wee HL. Current and future economic burden of diabetes among working-age adults in Asia: conservative estimates for Singapore from 2010-2050. BMC Public Health. 2016 Feb 16;16:153. doi: 10.1186/s12889-016-2827-1. PMID 26880337
- [Background] Roystonn K, Lau JH, AshaRani PV, Siva Kumar FD, Wang P, Sum CF, Lee ES, Chong SA, Subramaniam M. Recognition of diabetes and sociodemographic predictors: results of a cross-sectional nationwide population-based survey in Singapore. BMJ Open. 2022 Mar 1;12(3):e050425. doi: 10.1136/bmjopen-2021-050425. PMID 35232779
- [Background] Quah JH, Liu YP, Luo N, How CH, Tay EG. Younger adult type 2 diabetic patients have poorer glycaemic control: a cross-sectional study in a primary care setting in Singapore. BMC Endocr Disord. 2013 Jun 3;13:18. doi: 10.1186/1472-6823-13-18. PMID 23725198
- [Background] Lee CS, Tan JHM, Sankari U, Koh YLE, Tan NC. Assessing oral medication adherence among patients with type 2 diabetes mellitus treated with polytherapy in a developed Asian community: a cross-sectional study. BMJ Open. 2017 Sep 14;7(9):e016317. doi: 10.1136/bmjopen-2017-016317. PMID 28912194
- [Background] Tan KW, Dickens BSL, Cook AR. Projected burden of type 2 diabetes mellitus-related complications in Singapore until 2050: a Bayesian evidence synthesis. BMJ Open Diabetes Res Care. 2020 Mar;8(1):e000928. doi: 10.1136/bmjdrc-2019-000928. PMID 32184203
- [Background] Tan JK, Salim NNM, Lim GH, Chia SY, Thumboo J, Bee YM. Trends in diabetes-related complications in Singapore, 2013-2020: A registry-based study. PLoS One. 2022 Oct 11;17(10):e0275920. doi: 10.1371/journal.pone.0275920. eCollection 2022. PMID 36219616
- [Background] Rothman AJ, Kiviniemi MT. Treating people with information: an analysis and review of approaches to communicating health risk information. J Natl Cancer Inst Monogr. 1999;(25):44-51. doi: 10.1093/oxfordjournals.jncimonographs.a024207. PMID 10854457
- [Background] Roach P, Marrero D. A critical dialogue: communicating with type 2 diabetes patients about cardiovascular risk. Vasc Health Risk Manag. 2005;1(4):301-7. doi: 10.2147/vhrm.2005.1.4.301. PMID 17315602
- [Background] Paling J. Strategies to help patients understand risks. BMJ. 2003 Sep 27;327(7417):745-8. doi: 10.1136/bmj.327.7417.745. PMID 14512489
- [Background] Naik G, Ahmed H, Edwards AG. Communicating risk to patients and the public. Br J Gen Pract. 2012 Apr;62(597):213-6. doi: 10.3399/bjgp12X636236. No abstract available. PMID 22520906
- [Background] Gao R, Guo H, Liu Y, Pang Y, Zhang X, Lian X, Yu T, Zhu L, Li F. Effects of message framing on self-management behaviour among patients with type 2 diabetes: a randomised controlled trial protocol. BMJ Open. 2022 Jun 28;12(6):e056450. doi: 10.1136/bmjopen-2021-056450. PMID 35768085
- [Background] Garcia-Retamero R, Okan Y, Cokely ET. Using visual aids to improve communication of risks about health: a review. ScientificWorldJournal. 2012;2012:562637. doi: 10.1100/2012/562637. Epub 2012 May 2. PMID 22629146
- [Background] Trevena L. Assessing, communicating, and managing risk in general practice. Br J Gen Pract. 2014 Apr;64(621):166-7. doi: 10.3399/bjgp14X677725. No abstract available. PMID 24686863
- [Background] Welschen LM, Bot SD, Dekker JM, Timmermans DR, van der Weijden T, Nijpels G. The @RISK Study: Risk communication for patients with type 2 diabetes: design of a randomised controlled trial. BMC Public Health. 2010 Aug 5;10:457. doi: 10.1186/1471-2458-10-457. PMID 20687924
- [Background] Welschen LM, Bot SD, Kostense PJ, Dekker JM, Timmermans DR, van der Weijden T, Nijpels G. Effects of cardiovascular disease risk communication for patients with type 2 diabetes on risk perception in a randomized controlled trial: the @RISK study. Diabetes Care. 2012 Dec;35(12):2485-92. doi: 10.2337/dc11-2130. Epub 2012 Aug 24. PMID 22923669
- [Background] Rouyard T, Leal J, Baskerville R, Velardo C, Salvi D, Gray A. Nudging people with Type 2 diabetes towards better self-management through personalized risk communication: A pilot randomized controlled trial in primary care. Endocrinol Diabetes Metab. 2018 Jun 22;1(3):e00022. doi: 10.1002/edm2.22. eCollection 2018 Jul. PMID 30815556
- [Background] Mao L, Lu J, Zhang Q, Zhao Y, Chen G, Sun M, Chang F, Li X. Family-based intervention for patients with type 2 diabetes via WeChat in China: protocol for a randomized controlled trial. BMC Public Health. 2019 Apr 5;19(1):381. doi: 10.1186/s12889-019-6702-8. PMID 30953483
- [Background] Feng Y, Zhao Y, Mao L, Gu M, Yuan H, Lu J, Zhang Q, Zhao Q, Li X. The Effectiveness of an eHealth Family-Based Intervention Program in Patients With Uncontrolled Type 2 Diabetes Mellitus (T2DM) in the Community Via WeChat: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2023 Mar 20;11:e40420. doi: 10.2196/40420. PMID 36939825
- [Background] Fang HSA, Tan NC, Tan WY, Oei RW, Lee ML, Hsu W. Patient similarity analytics for explainable clinical risk prediction. BMC Med Inform Decis Mak. 2021 Jul 1;21(1):207. doi: 10.1186/s12911-021-01566-y. PMID 34210320
- [Background] Oei RW, Fang HSA, Tan WY, Hsu W, Lee ML, Tan NC. Using Domain Knowledge and Data-Driven Insights for Patient Similarity Analytics. J Pers Med. 2021 Jul 22;11(8):699. doi: 10.3390/jpm11080699. PMID 34442343
- [Background] Stefanut AM, Vintila M. Psychotherapeutic intervention on breast self-examination based on Health Belief Model. Curr Psychol. 2022 Feb 21:1-9. doi: 10.1007/s12144-022-02871-z. Online ahead of print. PMID 35221635
- [Background] Walrave M, Waeterloos C, Ponnet K. Adoption of a Contact Tracing App for Containing COVID-19: A Health Belief Model Approach. JMIR Public Health Surveill. 2020 Sep 1;6(3):e20572. doi: 10.2196/20572. PMID 32755882
- [Background] Robinson CA. Trust, Health Care Relationships, and Chronic Illness: A Theoretical Coalescence. Glob Qual Nurs Res. 2016 Aug 12;3:2333393616664823. doi: 10.1177/2333393616664823. eCollection 2016 Jan-Dec. PMID 28508016
- [Background] Gorawara-Bhat R, Huang ES, Chin MH. Communicating with older diabetes patients: self-management and social comparison. Patient Educ Couns. 2008 Sep;72(3):411-7. doi: 10.1016/j.pec.2008.05.011. Epub 2008 Jul 18. PMID 18639997
- [Background] Lim DYZ, Chia SY, Abdul Kadir H, Mohamed Salim NN, Bee YM. Establishment of the SingHealth Diabetes Registry. Clin Epidemiol. 2021 Mar 16;13:215-223. doi: 10.2147/CLEP.S300663. eCollection 2021. PMID 33762850
- [Background] Gibbons FX, Buunk BP. Individual differences in social comparison: development of a scale of social comparison orientation. J Pers Soc Psychol. 1999 Jan;76(1):129-42. doi: 10.1037//0022-3514.76.1.129. PMID 9972558
- [Background] Chan AHY, Horne R, Hankins M, Chisari C. The Medication Adherence Report Scale: A measurement tool for eliciting patients' reports of nonadherence. Br J Clin Pharmacol. 2020 Jul;86(7):1281-1288. doi: 10.1111/bcp.14193. Epub 2020 May 18. PMID 31823381
- [Background] Toobert DJ, Hampson SE, Glasgow RE. The summary of diabetes self-care activities measure: results from 7 studies and a revised scale. Diabetes Care. 2000 Jul;23(7):943-50. doi: 10.2337/diacare.23.7.943. PMID 10895844